CLINICAL TRIAL: NCT01377103
Title: Cardiovascular and Functional Effects of Testosterone Therapy for Hypogonadal Patients With Heart Failure
Brief Title: Testosterone Therapy in Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Ernst Schwarz, MD, PhD, Affiliate, Cedars-Sinai Heart Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TT-1
Record Dates: First submitted 2011-05-18; First posted 2011-06-21 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2011-04

CONDITIONS: Heart Failure; Hypogonadism
Keywords: heart failure; hypogonadism; testosterone
MeSH Terms: conditions — Heart Failure; Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Gel
  Interventions: Drug: Placebo
- Testosterone Supplementation (Active Comparator): Testosterone Gel
  Interventions: Drug: testerone gel

INTERVENTIONS:
Drug: testerone gel — 5g daily for 4 weeks then 7.5 or 10g daily for 8 weeks; transdermal testosterone gel
  Other Names: AndroGel(R)
  Arms: Testosterone Supplementation
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether benefits of topical testosterone on symptoms and function of male HF patients, and its effects on rehospitalization rates and quality of life.

DETAILED DESCRIPTION:
Recent evidence has started to emerge regarding the benefits of testosterone in the heart failure (HF) population. Firstly, testosterone directly augments vascular resistance by causing vasodilation of peripheral vessels which can decrease afterload and improve cardiac output. In addition, testosterone causes coronary artery vasodilation and improves cardiac ischemic threshold based on subjective and objective measures. Clinically, several studies have pointed out the potential benefits patients with HF can derive from testosterone therapy. Measures of cardiopulmonary function tests, six minute walk test, incremental shuttle walk test and baroreflex sensitivity, all of which have prognostic implications for patients with HF, show improvement with the addition of testosterone therapy to traditional-medical management. In addition to these objective measurements, mood, NYHA functional class and muscle strength are all improved by treatment with testosterone supplementation. While past studies have used functional and prognostic measures as outcomes, other issues common in patients with HF, such as sexual dysfunction and repeat hospitalizations, have the potential for improvement with testosterone therapy

The majority of studies performed in the past have utilized intramuscular or transdermal patch delivery systems of testosterone as a means for supplementation. These methods have inherent issues as a means of treatment as patients often times do not have the means to receive intramuscular injections and patches have a high level of skin reactions making compliance difficult. Topical administration of testosterone gel may prove to be a more efficacious method for testosterone supplementation with a lower side effect profile and adequate absorption. It has been used with success by the general public for treatment of hypogonadal symptoms, but has not been studied in the HF population. With the emergence of studies showing promising benefits of testosterone supplementation in the HF population, the ease of topical administration for this population would provide benefits to millions suffering from HF.

The investigators study aims to find the benefits of topical testosterone on symptoms and function of HF patients, and its effects on rehospitalization rates and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* male
* NYHA class II-IV Heart Failure
* age > 35 < 80
* total testosterone level of <5 ng/ml

Exclusion Criteria:

* elevated prostate specific antigen
* elevated total or free testosterone level
* prostate cancer or evidence of symptomatic prostatism
* untreated prolactinemia or history of breast cancer

Ages: 36 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
heart failure outcomes | 16 months
  rehospitalization rates, mortality, New York Heart Association class and symptomatolgy
depression and mood | 16 months
  Beck Depression Inventory: a 21-question multiple-choice self-report inventory for measuring the severity of depression
quality of life | 16 months
  Minnesota Living with Heart Failure Questionnaire

SECONDARY OUTCOMES:
overall satisfaction | 16 months
  Minnesota Living with Heart Failure Questionnaire
compliance | 16 months
  documentation of study medication usage
markers for heart failure | 16 months
  natriuretic peptide, creatinine, and left ventricular ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Schwarz, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center